CLINICAL TRIAL: NCT00667732
Title: Metformin, Exenatide, and Glargine Insulin in Combination for Treatment of Patients With Type 2 Diabetes
Brief Title: How Glargine Insulin, Oral Diabetes Medications and Exenatide May Improve Blood Sugar Control and Weight Gain in Type 2 Diabetics
Acronym: MEXELIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Matthew C. Riddle, Matthew Riddle, MD, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IND 75,235
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; insulin; byetta; glucose; blood sugar; metformin; A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive exenatide as part of their diabetes treatment
  Interventions: Drug: exenatide
- 2 (Placebo Comparator): Participants will receive placebo rather than exenatide as part of their diabetes treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — 5mcg twice a day, increasing to 10mcg twice a day for 24 weeks
  Other Names: Byetta
  Arms: 1
Drug: placebo — 5mcg twice a day, increased to 10mcg twice a day for 24 weeks
  Arms: 2

SUMMARY:
This study is designed to look at how using glargine insulin with oral diabetes medications and exenatide may improve control of blood sugar levels and weight gain in type 2 diabetics.

The main study will last 32 weeks. However, all participants completing 32 weeks will be invited to continue for another 24 weeks taking the insulin and oral medication and exenatide treatment. This extension comparing insulin and oral medication with insulin and oral medication and exenatide will look at the long term weight loss/gain and blood sugar level control effects of this new drug regimen.

There is also a sub-study in the Clinical Research Center (CRC), which requires two 38-hour inpatient stays during the main study. This study offers the opportunity to study 24-hour blood sugar and metabolic patterns quantitatively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with type 2 diabetes
* Taking metformin at least 1000 mg daily plus a secretagogue, an alpha glucosidase inhibitor, a thiazolidinedione, or a single injection of any kind of insulin up to 0.4 units/kg daily for > 3 months
* Age range 30 to 70 years
* Body mass index 25-45 kg/m2
* HbA1c 7.0 to 10.0% (or 7.0 to 8.5% if the second antihyperglycemic agent is insulin)
* Less than 50% of randomized participants will have used insulin previously

Exclusion Criteria:

* Use of more than two antihyperglycemic agents within the last 3 months
* Use of more than one daily injection of any kind of insulin in the last 3 months
* Positive anti-GAD antibody (test required in screening)
* Fasting C-peptide <0.5 ng/mL (test required in screening)
* Pregnancy (test required in screening if able to conceive) or lactation
* Excessive use of alcohol or evidence of other form of drug dependency
* Unwillingness or inability to grant informed consent
* Unwillingness or inability to perform self-monitoring of blood glucose
* Unwillingness or inability to inject insulin and/or inject exenatide
* Serum creatinine >1.3 mg/dL in women or 1.4 in men
* Retinopathy which has required photocoagulation for treatment
* Major active systemic illness (e.g. neoplastic disorder, symptomatic ischemic heart disease, congestive heart failure) that might interfere with performing the study protocol
* Clinically significant gastrointestinal disorder including prior gastric or intestinal surgery for weight-control
* Ongoing use of any drug (e.g. narcotic analgesic, tricyclic antidepressant) that might alter gastric emptying
* Use prednisone or other systemic glucocorticoid drug in the last 3 months
* Use of any drug for weight-control (e.g. sibutramine, phentermine, orlistat) in the last 3 months
* Use of any unproven investigational drug within the last 3 months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Riddle, MD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Medstar Research Institute, Washington D.C., District of Columbia
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Health and Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: March 2007 - February 2009 Participant source: medical clinics, local communities
Pre-assignment Details: There were 8 weeks of open-label exenatide use before enrollment into the randomized portion of the study to ensure patients ability to tolerate medication before adding insulin to the medication regimen.
Groups:
- Run-In Group: All participants took exenatide twice daily in addition to their Metformin dose.
  A subset of participants agreed to a substudy (20 pts) and had a glucose and metabolic profile done at this time.
- Exenatide Group: After run-in participants were randomized to exenatide.
  exenatide : 5mcg twice a day, increasing to 10mcg twice a day for 24 weeks
  metformin: continued at same dose participant entered study on.
  Lantus Insulin: titrated per protocol depending on blood sugar levels
  In extension period, participants continued regular regimen with open label exenatide
- Placebo Group: After run-in participants were randomized to placebo.
  placebo : 5mcg twice a day, increased to 10mcg twice a day for 24 weeks
  metformin: continued at same dose participant entered study on.
  Lantus Insulin: titrated per protocol depending on blood sugar levels
  In extension period, participants continued regular regimen with open label exenatide instead of placebo
Period: Run -In (8 Weeks)
Arm/Group | Run-In Group | Exenatide Group | Placebo Group
Started | 41 | 0 | 0
Participants Enrolled in Substudy | 20 | 0 | 0
Completed | 34 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Period: Randomization (24 Weeks)
Arm/Group | Run-In Group | Exenatide Group | Placebo Group
Started | 0 | 17 | 17
Participants Enrolled in Substudy | 0 | 11 | 9
Completed | 0 | 16 | 17
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Extension (26 Weeks)
Arm/Group | Run-In Group | Exenatide Group | Placebo Group
Started | 0 | 14 | 17
Completed | 0 | 14 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exenatide Group: Participants will receive exenatide as part of their diabetes treatment
  exenatide : 5mcg twice a day, increasing to 10mcg twice a day for 24 weeks
- Placebo Group: Participants will receive placebo rather than exenatide as part of their diabetes treatment
  placebo : 5mcg twice a day, increased to 10mcg twice a day for 24 weeks
- Total: Total of all reporting groups
Arm/Group | Exenatide Group | Placebo Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Intent to Treat Participants Randomized and Treated in Each Arm Who Had Lab-measured A1c <6.5% at 24 Weeks of Treatment
Time Frame: After 24 weeks of randomized treatment
Population: Intent to treat. All participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Group | Placebo Group
Number analyzed (Participants) | 17 | 17
percentage of participants | 47 [5.7 to 9.3] | 12 [5.7 to 9.8]

2. Secondary Outcome: The Percentage of Per Protocol Participants Randomized and Treated in Each Arm Who Had Lab-measured A1c <6.5% at 24 Weeks of Treatment
Description: efficacy criteria, 50% of per protocol participants reached A1c target of <6.5%
Time Frame: After 24 weeks of randomized treatment
Population: Per protocol, all participants who completed treatment
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Group | Placebo Group
Number analyzed (Participants) | 16 | 17
percentage of participants | 50 (0.27) | 12

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the screening visit to final clinic visit totaling 59 weeks.
Description: All participants who received at least one dose of treatment during appropriate period
Groups:
- Run-In Group: All participants took exenatide twice daily in addition to their Metformin dose.
- Exenatide Randomization Group: After run-in participants were randomized to exenatide. exenatide : 5mcg twice a day, increasing to 10mcg twice a day for 24 weeks metformin: continued at same dose participant entered study on. Lantus Insulin: titrated per protocol depending on blood sugar levels
- Placebo Randomization Period: After run-in participants were randomized to placebo. placebo : 5mcg twice a day, increased to 10mcg twice a day for 24 weeks metformin: continued at same dose participant entered study on. Lantus Insulin: titrated per protocol depending on blood sugar levels
- Exenatide Open-Label (Previous Exenatide): Participants who were in the Exenatide Arm during randomization who received open label: exenatide : 5mcg twice a day, increasing to 10mcg twice a day for 24 weeks metformin: continued at same dose participant entered study on. Lantus Insulin: titrated per protocol depending on blood sugar level
- Exenatide Open-Label (Previous Placebo): Participants who were in the Placebo Arm during randomization who received open label: exenatide : 5mcg twice a day, increasing to 10mcg twice a day for 24 weeks metformin: continued at same dose participant entered study on. Lantus Insulin: titrated per protocol depending on blood sugar level
Arm/Group | Run-In Group | Exenatide Randomization Group | Placebo Randomization Period | Exenatide Open-Label (Previous Exenatide) | Exenatide Open-Label (Previous Placebo)
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/17 | 0/17 | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 21/38 | 15/17 | 10/17 | 11/14 | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Group (N=38) | Exenatide Randomization Group (N=17) | Placebo Randomization Period (N=17) | Exenatide Open-Label (Previous Exenatide) (N=14) | Exenatide Open-Label (Previous Placebo) (N=17)
Nausea (Gastrointestinal disorders) | 13 | 3 | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 4 | 1 | 1 | 1 | 1
Stomach ache, upset (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0
Heartburn, reflux (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0
diarrhea, loose stools (Gastrointestinal disorders) | 3 | 2 | 0 | 3 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 4 | 3 | 3 | 2
Headache (Nervous system disorders) | 3 | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Hiatal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Sour Taste (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dental Work (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis, stomach flu (Gastrointestinal disorders) | 0 | 2 | 4 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Allergies (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Strep Throat (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Left wrist sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Left 5th toe fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall with bruised arm, leg (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Right Ankle Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Right thumb pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Left foot pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Right and left shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Right ankle swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
left toe swelling (gout) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Left wrist pain and numbness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Elevated Creatinine (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Lost voice (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Injection site redness, itching (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Left wrist pigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Conjunctival hemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0
Dry Eyes (Eye disorders) | 0 | 0 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Decreased energy (General disorders) | 0 | 0 | 0 | 0 | 1
Cold/flu (Infections and infestations) | 0 | 0 | 0 | 4 | 3
Sore Throat (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lymph node enlargement, cervical (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paronychial infection, finger (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cold sore, lip (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ankle sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Motor vehicle accident with facial laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Rib Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthritis, leg (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Aching elbows (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Bell's Palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Numbness, arms, hands (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Carpal Tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ulnar neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Endocrine disorders) | 0 | 10 | 8 | 8 | 10
Fall with leg contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less